CLINICAL TRIAL: NCT06420219
Title: An Integrative Multi-Omic Characterization of Head and Neck Carcinogenesis, Progression and Recurrence
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 7H-23-4; NCI-2024-01559 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7H-23-4 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2024-03-25; First posted 2024-05-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo photography, blood sample collection, tissue collection and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the cell and biomarkers associated with the aggressive behavior of cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. High-resolution single-cell profiling of Cancer-associated fibroblasts (CAFs) in Human papillomavirus (HPV)+ Oropharyngeal Squamous Cell Carcinoma (OPSCC) and metastatic lymph nodes.

OUTLINE: This is an observational study.

Patients undergo photography, blood sample collection, tissue collection and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis/disease status: New diagnosis of head and neck cancer
* Allowable type and amount of prior therapy: No prior treatment
* Age ≥ 18 years.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients who have had treatment of head and neck cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a new diagnosis of head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2028-03-25 (Estimated); Study Completion 2029-03-25 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years
Disease free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Albert Y Han, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States